CLINICAL TRIAL: NCT01904747
Title: A Phase 1, Open-Label 4 Sequence 4 Period Crossover Study Of Palbociclib (PD-0332991) In Healthy Volunteers To Estimate The Effect Of Food On The Bioavailability Of Palbociclib
Brief Title: Characterization Of The Effect Of Food On Palbociclib (PD-0332991) Absorption
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A5481021
Record Dates: First submitted 2013-07-01; First posted 2013-07-22 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Healthy
Keywords: Food; Bioavailability; Fasted; Fed
MeSH Terms: conditions — Lecithin Cholesterol Acyltransferase Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Palbociclib given to healthy volunteers (Experimental)
  Interventions: Drug: Palbociclib administered Fasted; Drug: Palbociclib administered Fed high calorie; Drug: Palbociclib administered Fed low calorie; Drug: Palbociclib administered Fed moderate calorie

INTERVENTIONS:
Drug: Palbociclib administered Fasted — palbociclib given under fasting 10 hrs overnight; capsule form, 125 mg single dose
Drug: Palbociclib administered Fed high calorie — palbociclib given right after a high fat high calorie meal; capsule form, 125 mg single dose
Drug: Palbociclib administered Fed low calorie — palbociclib given right after a low fat low calorie meal; capsule form, 125 mg single dose
Drug: Palbociclib administered Fed moderate calorie — palbociclib given between moderate calorie meal; capsule form, 125 mg single dose

SUMMARY:
This study is intended to quantify the effect of food on the extent of absorption of palbociclib.

The caloric content of the food and the time of the meals with respect to palbociclib administration may influence the capacity of the body to absorb the drug.

High and low calorie meals will be given to the subjects 30 minutes before palbociclib administration as 2 of the 3 conditions to compare with completely absence of food in the body when dosing (fasted).The third condition to test and compare with fasted stage will be the administration of food before and after palbociclib administration.

This information will help the program to decide wether or not the presence of food when dosing palbociclib help with its absorption and to what extent it does help. Based on the collected information, a recommendation about the administration of palbociclib with food will be provided to patients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects and/or female subjects of non-childbearing potential between the ages of 18 and 55 years
* Evidence of a personally signed and dated informed consent document indicating that the subject (or a legal representative) has been informed of all pertinent aspects of the study
* Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease
* Any condition possibly affecting drug absorption
* Male subjects who are unwilling or unable to use a highly effective method of contraception

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2013-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] | 144 hrs
  AUC (0 - 8)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - 8). It is obtained from AUC (0 - t) plus AUC (t - 8).
Maximum Observed Plasma Concentration (Cmax) | 144 hrs

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 144 hrs
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)] | 144 hrs
  AUC (0-t)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-t)
Area under the Concentration-Time Curve (AUC) from 0 to 72 hrs | 144 hrs
  AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption.
Apparent Oral Clearance (CL/F) | 144 hrs
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 144 hrs
Apparent Volume of Distribution (Vz/F) | 144 hrs
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Plasma Decay Half-Life (t1/2) | 144 hrs
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Ruiz-Garcia A, Plotka A, O'Gorman M, Wang DD. Effect of food on the bioavailability of palbociclib. Cancer Chemother Pharmacol. 2017 Mar;79(3):527-533. doi: 10.1007/s00280-017-3246-4. Epub 2017 Feb 15. PMID 28204912
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5481021&StudyName=Characterization%20Of%20The%20Effect%20Of%20Food%20On%20Palbociclib%20%28PD-0332991%29%20Absorption%0A